CLINICAL TRIAL: NCT04711629
Title: Clinical Characteristics of Chronic Obstructive Pulmonary Patients Who Continue to Smoke
Brief Title: Clinical Features of Smoker Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IKCU-INAZ
Record Dates: First submitted 2020-11-05; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Copd; Smoking
Keywords: copd; smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Intervention Model Description: Smoker COPD Ex Smoker COPD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoker COPD (Experimental): Patients who continue to smoke
  Interventions: Other: Clinical Tests
- Ex-smoker COPD (Active Comparator): Patients who quit smoking.
  Interventions: Other: Clinical Tests

INTERVENTIONS:
Other: Clinical Tests — Respiratory function test, arterial blood gas analysis, six-minute walking test (6-MWT), mMRC Dyspnea Scale, St George Quality of Life Questionnaire and Hospital Anxiety Depression Scale

SUMMARY:
Smoking is the most important factor in the etiology of COPD. Some of the patients with COPD continue to smoke despite knowing this situation or they cannot quit even if they want.

The aim of this study is; To examine patients with COPD who continue to smoke in terms of perception of dyspnea, exercise capacity, psychological symptoms and quality of life.

DETAILED DESCRIPTION:
The study was designed prospectively. Patients with COPD who apply to the pulmonary rehabilitation outpatient clinic will be included.

The data of patients with COPD who are eligible for PR and have been pre-evaluated will be scanned. Respiratory function test, arterial blood gas analysis, six-minute walking test (6-MWT), mMRC Dyspnea Scale, St George Quality of Life Questionnaire and Hospital Anxiety Depression Scale will be used in the study. Patients with COPD who smoke will constitute the study group, and those who quit smoking will constitute the control group.

ELIGIBILITY:
Inclusion Criteria:

* Smoker COPD Patients who smoker

Exclusion Criteria:

* Not volunteer to participate the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | 6 minutes
  Six minutes walk test

SECONDARY OUTCOMES:
Respiratory Functions | 30 minutes
  Pulmonary Function Test Pulmonary function test (PFT) which is noninvasive tests that show how well the lungs are working. The tests will measure FEV1; It is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
  FVC: It s the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry FEV1/FVC: It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Dyspnea Sensation | 20 minutes
  Modified Medical Research Council (MMRC)" dyspnea scale, which consists of 5 items ranging between 1 and 5, to determine the severity of patients' shortness of breath.
Disease Specific Quality of Life | 20 minutes
  St. George's Respiratory Questionnaire (SGRQ) to determine disease-specific quality of life. At this scale, high scores define worsened disease and increased symptoms.
Anxiety | 20 minutes
  Hospital Anxiety and Depression (HAD) Inventory for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.
Depression | 20 minutes
  Hospital Anxiety and Depression (HAD) Inventory for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.
Body Mass Index | 5 minutes
  Body mass index is calculated by dividing body mass by the square of length in meters.

IPD SHARING:
Plan to Share IPD: No